CLINICAL TRIAL: NCT00362219
Title: Topical Morphine for Analgesia in Patients With Skin Grafts
Status: Withdrawn | Phase: Phase 3 | Type: Interventional
Why Stopped: no patients were recrueted
Sponsor: Rambam Health Care Campus (Other)
Responsible Party: Principal Investigator, Yehuda Ullmann MD, Head, Plastic Surgery Department, Rambam Health Care Campus
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: RMC-2468.CTIL
Record Dates: First submitted 2006-08-08; First posted 2006-08-09 (Estimated); Last update posted 2022-05-03 (Actual); Status verified 2022-04

CONDITIONS: Skin Transplantation; Pain
Keywords: topical; morphine; pain; skin-wound; skin-graft; peripheral analgesia; burn
MeSH Terms: conditions — Pain; Burns | interventions — Morphine

STUDY DESIGN:
Who Masked: Participant, Care Provider, Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (4):
- Placebo (Placebo Comparator): Gel with no active ingredient
  Interventions: Other: Placebo
- Morphine .25 mg (Active Comparator): Gel with 0.25 mg morphine per 100cm2 square of wound
  Interventions: Drug: Morphine - .25 mg
- Morphine - .75 mg. (Active Comparator): Gel with 0.75 mg morphine per 100cm2 square of wound.
  Interventions: Drug: Morphine
- Morphine 1.25 mg. (Active Comparator): Gel with 1.25 mg morphine per 100cm2 square of wound.
  Interventions: Drug: Morphine

INTERVENTIONS:
Other: Placebo — Gel with no active ingredient.
  Arms: Placebo
Drug: Morphine - .25 mg — gel with 0.25 mg morphine per 100cm2 square of wound.
  Arms: Morphine .25 mg
Drug: Morphine — Gel with 0.75 mg morphine per 100cm2 square of wound.
  Arms: Morphine - .75 mg.
Drug: Morphine — Gel with 1.25 mg morphine per 100cm2 square of wound.
  Arms: Morphine 1.25 mg.

SUMMARY:
The management of pain endured by patients after skin grafting is complex. Pain is the single most distressing symptom but as it is difficult to manage, it is often under-treated. These patients may experience pain from two types of wound: the original injury and from "skin-donor" sites, areas of healthy skin from which skin is surgically removed and used to cover the original injury. As the section of skin which is removed is standardized, the wound created at the donor site is uniform and so provides a model of an acute wound.

Opioids (such as morphine) are the backbone of treating the moderate to severe pain experienced by any patient. But due to their potentially severe side effects and that some patients do not experience sufficient relief from the treatment, optimal treatment schedules are still being sought after.

Topically applied morphine has provided effective and safe analgesia in several clinical models. We, therefore, wish to apply this treatment modality onto skin-graft donor wounds. If found to be effective this could be an appealing non-invasive method to treat the pain of this type of wound.

DETAILED DESCRIPTION:
Administration of morphine into the knee joint is the best-studied clinical procedure documenting the use of topically-applied opioids. When 1-5 mg morphine were injected into the knee joint, patients experienced pain relief for up to 24 hours, whereas similar doses given systemically (i.e. intravenously) were effective for 2-4 hours. Furthermore, the analgesic effect was reversed when the opioid antagonist naloxone was injected into the knee joint. Both these findings indicate that the effect is mediated by local opioid receptors in the knee joint.

Peripheral analgesic effects of opioids are not detectable in normal tissue but appear minutes to hours after initiation of inflammation. This suggests that opioid receptors are already present in the peripheral nerve terminals but under normal conditions they are not functional.

Research on application of opioids to skin wounds is very sparse and has primarily been performed in palliative care patients. These reports demonstrate that topical opioid gel (morphine or diamorphine) provided rapid and effective relief. In some patients pain subsided within 20 minutes after application with a long-lasting (7-8 hours) effect. Fundamental aspects regarding topical application of opioids onto skin wounds are still lacking. For example, issues such as optimal dose and dose-effect relationships have not been investigated. We hope to determine these in this study.

ELIGIBILITY:
Inclusion Criteria:

* Patients undergoing skin-grafting
* American Society of Anesthesiologists (ASA) classification I-II
* Written consent
* Either sex
* Able to self-asses and report their pain level

Exclusion Criteria:

* Alcohol abuse or addiction - current
* Opioids and benzodiazepines abuse - life time
* Known hypersensitivity to morphine
* Major renal or hepatic dysfunction
* Pregnancy or lactation
* Sleep-apnoea-syndrome
* Diabetes
* Participation in other clinical studies

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2022-01 (Estimated); Primary Completion 2023-12 (Estimated); Study Completion 2024-12 (Estimated)

PRIMARY OUTCOMES:
Pain score in first 24 hours | 24 hours after application of the medication
  Sum of the differences in pain scores between the skin-donor site vs. original injury site taken over a 24 hour period after application of the medication.

SECONDARY OUTCOMES:
Pain Score | 24 hours after surgery
  Pain score at skin-donor site using an abbreviated form of the McGill Pain Questionnaire
Time course of analgesia for each drug concentration | First 24 hours after surgery
  Time course of analgesia for each drug concentration
Side effects | First 24 hours after surgery
  Presence and severity of side effects: (a) central (nausea, vomiting, sedation, purities) and (b) local (burning, tingling, wheal, flare)
Supplementary analgesic medications | First 24 hours after surgery
  Concurrent, supplementary, "rescue", analgesic medication (i.v.or oral morphine), given during the first 24 hours post operatively
Analgesic medicine from 2nd post-operative day until dressings are removed. | Day 2 post-surgery through 12th post-op day on average
  Analgesic medication (type and dose), given from the second post-operative day until dressings are removed for the first time (= the 12th post-operataive day, on average).
Pain score collection | Twice daily from day 2 post-op until day 8 post-op
  Pain scores at donor and original injury, twice daily, from the second post-operative day until dressings are removed for the first time - up until 8th post-op day
Wound assessment | Average day 12 post-operative
  Assessment of the wound once the dressings are removed

CONTACTS AND LOCATIONS:
Overall Officials: Yehuda Ullman, M.D., Principal Investigator — Rambam Health Care Campus
Locations (1):
- Department of Plastic Surgery, Rambam Medical Center, Haifa, Israel

REFERENCES:
- [Background] Krajnik M, Zylicz Z, Finlay I, Luczak J, van Sorge AA. Potential uses of topical opioids in palliative care--report of 6 cases. Pain. 1999 Mar;80(1-2):121-5. doi: 10.1016/s0304-3959(98)00211-5. PMID 10204724
- [Background] Stein C, Comisel K, Haimerl E, Yassouridis A, Lehrberger K, Herz A, Peter K. Analgesic effect of intraarticular morphine after arthroscopic knee surgery. N Engl J Med. 1991 Oct 17;325(16):1123-6. doi: 10.1056/NEJM199110173251602. PMID 1653901
- [Background] Porzio G, Aielli F, Verna L, Cannita K, Marchetti P, Ficorella C. Topical morphine in the treatment of painful ulcers. J Pain Symptom Manage. 2005 Oct;30(4):304-5. doi: 10.1016/j.jpainsymman.2005.08.011. No abstract available. PMID 16256893
- [Background] Ribeiro MD, Joel SP, Zeppetella G. The bioavailability of morphine applied topically to cutaneous ulcers. J Pain Symptom Manage. 2004 May;27(5):434-9. doi: 10.1016/j.jpainsymman.2003.09.011. PMID 15120772
- [Background] Stein A, Yassouridis A, Szopko C, Helmke K, Stein C. Intraarticular morphine versus dexamethasone in chronic arthritis. Pain. 1999 Dec;83(3):525-532. doi: 10.1016/S0304-3959(99)00156-6. PMID 10568861
- [Background] Zeppetella G, Ribeiro MD. Morphine in intrasite gel applied topically to painful ulcers. J Pain Symptom Manage. 2005 Feb;29(2):118-9. doi: 10.1016/j.jpainsymman.2004.12.006. No abstract available. PMID 15733803
- [Background] Stein C, Schafer M, Machelska H. Attacking pain at its source: new perspectives on opioids. Nat Med. 2003 Aug;9(8):1003-8. doi: 10.1038/nm908. PMID 12894165